CLINICAL TRIAL: NCT00412958
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Masked, Parallel Group, Dose-Ranging Clinical Trial of Intravitreal Microplasmin in Patients Undergoing Surgical Vitrectomy: The MIVI III (Microplasmin For Vitreous Injection III) Trial
Brief Title: A Study of the Safety and Efficacy of Microplasmin to Induce a Posterior Vitreous Detachment (MIVI III)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-MV-003
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-04

CONDITIONS: Vitrectomy
MeSH Terms: interventions — microplasmin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ocriplasmin 25µg (Experimental): 25µg of ocriplasmin intravitreal injection
  Interventions: Drug: Ocriplasmin 25µg
- Ocriplasmin 75µg (Experimental): 75µg of ocriplasmin intravitreal injection
  Interventions: Drug: Ocriplasmin 75µg
- Ocriplasmin 125µg (Experimental): 125µg of ocriplasmin intravitreal injection
  Interventions: Drug: Ocriplasmin 125µg
- Placebo (Placebo Comparator): Intravitreal injection of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ocriplasmin 25µg — Intravitreal injection of 0.1 ml of ocriplasmin solution containing 25µg of ocriplasmin.
  Other Names: Microplasmin
  Arms: Ocriplasmin 25µg
Drug: Ocriplasmin 75µg — Intravitreal injection of 0.1 ml of ocriplasmin solution containing 75µg of ocriplasmin.
  Other Names: Microplasmin
  Arms: Ocriplasmin 75µg
Drug: Ocriplasmin 125µg — Intravitreal injection of 0.1 ml of ocriplasmin solution containing 125µg of ocriplasmin.
  Other Names: Microplasmin
  Arms: Ocriplasmin 125µg
Drug: Placebo — Intravitreal injection of placebo
  Arms: Placebo

SUMMARY:
A multicenter study to compare multiple doses of intravitreal microplasmin in patients undergoing surgical vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom vitrectomy is indicated

Exclusion Criteria:

* Posterior Vitreous Detachment (PVD) present at baseline
* Vitreous hemorrhage
* Certain vitreoretinal conditions including proliferative disease, rhegmatogenous retinal detachment, and proliferative vitreoretinopathy (PVR)
* Have had a vitrectomy in the study eye at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2006-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Retina Centers, P.C., Tucson, Arizona
  - VMR Institute, Huntington Beach, California
  - Jules Stein Eye Institute/UCLA, Los Angeles, California
  - Retinal Consultants of San Diego, Poway, California
  - Retinal Consultants Medical Group, Sacramento, California
  - National Ophtlamic Research Institute, Fort Meyers, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Rush University Med. Ctr, Chicago, Illinois
  - Mailing add: New England Eye Center - Tufts, Boston, Massachusetts
  - Associated Retinal Consultants, P.C., Royal Oak, Michigan
  - Vitroretinal Surgery, PA, Minneapolis, Minnesota
  - Retina Vitreous Centre, PA, New Brunswick, New Jersey
  - Columbia University - Harkness Eye Institute, New York, New York
  - Retina Vitreous Surgeons of Central NY, New York, New York
  - Duke Eye Center, Durham, North Carolina
  - Retina Association of Cleveland, Lakewood, Ohio
  - Allegheny Ophthalmic & Orbital Associates, P.C., Pittsburgh, Pennsylvania
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Vitreoretinal Consultants, Houston, Texas
  - Valley Retina Institute, P.A., McAllen, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was recruited on 29 Mar 2007 and the last patient completed the study on 02 Oct 2008.
Groups:
- Ocriplasmin 25µg: 25µg ocriplasmin intravitreal injection.
- Ocriplasmin 75µg: 75µg ocriplasmin intravitreal injection.
- Ocriplasmin 125µg: 125µg ocriplasmin intravitreal injection.
Period: Overall Study
Arm/Group | Ocriplasmin 25µg | Ocriplasmin 75µg | Ocriplasmin 125µg | Placebo
Started | 29 | 33 | 32 | 31
Completed | 26 | 29 | 32 | 30
Not Completed | 3 | 4 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Transport issue | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ocriplasmin 25µg | Ocriplasmin 75µg | Ocriplasmin 125µg | Placebo | Total
Number analyzed (Participants) | 29 | 33 | 32 | 31 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (8.28) | 68.8 (9.07) | 66.9 (11.40) | 65.7 (11.60) | 66.1 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 20 | 22 | 85
  Male | 9 | 10 | 12 | 9 | 40

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving Total Posterior Vitreous Detachment (PVD) Without Creation of an Anatomical Defect
Description: The primary efficacy endpoint was the proportion of patients achieving total PVD without creation of an anatomical defect (ie, retinal hole, retinal detachment) based on surgeon visualization at the beginning of vitrectomy prior to suction or any other mechanical intervention.
Time Frame: Day 7
Population: Intent-To-Treat (ITT). Full Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | Ocriplasmin 25µg | Ocriplasmin 75µg | Ocriplasmin 125µg | Placebo
Number analyzed (Participants) | 29 | 33 | 32 | 30
percentage of participants | 13.8 | 18.2 | 31.3 | 10
Statistical Analysis 1: Comparison: Ocriplasmin 25µg vs Placebo; P-values are from Wald chi-square tests from a logistic regression model with study center and treatment as categorical fixed effects comparing active treatment groups with the placebo group as the reference group; Test type: Superiority or Other; p = 0.796, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.24 to 6.36]
Statistical Analysis 2: Comparison: Ocriplasmin 75µg vs Placebo; P-values are from Wald chi-square test from a logistic regression model with study center and treatment as categorical fixed effects comparing active treatment groups with the placebo group as the reference group; Test type: Superiority or Other; p = 0.447, Regression, Logistic; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.39 to 8.36]
Statistical Analysis 3: Comparison: Ocriplasmin 125µg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.107, Regression, Logistic; Odds Ratio (OR) = 3.28, 95% CI 2-sided [0.77 to 13.95]

ADVERSE EVENTS:
Time Frame: Adverse Events(AEs)/Serious Adverse Events(SAEs) were collected from injection day up to Day 180 post-injection.
Description: AEs/SAEs were assessed by the investigator at all study visits.
Arm/Group | Ocriplasmin 25µg | Ocriplasmin 75µg | Ocriplasmin 125µg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/29 | 3/33 | 0/32 | 2/31
Other Adverse Events (participants affected / at risk) | 29/29 | 32/33 | 31/32 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin 25µg (N=29) | Ocriplasmin 75µg (N=33) | Ocriplasmin 125µg (N=32) | Placebo (N=31)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinutis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anterior chamber inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bening pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin 25µg (N=29) | Ocriplasmin 75µg (N=33) | Ocriplasmin 125µg (N=32) | Placebo (N=31)
Conjunctival haemorrahge (Eye disorders) | 14 (17) | 18 (22) | 17 (18) | 22 (22)
Anterior chamber cell (Eye disorders) | 12 (13) | 13 (17) | 13 (16) | 7 (8)
Anterior chamber flare (Eye disorders) | 6 (6) | 7 (9) | 11 (12) | 6 (6)
Cataract nuclear (Eye disorders) | 9 (13) | 7 (8) | 8 (9) | 8 (12)
Macular oedema (Eye disorders) | 5 (6) | 10 (11) | 4 (4) | 7 (8)
Cataract (Eye disorders) | 6 (6) | 9 (9) | 7 (9) | 5 (5)
Eye pain (Eye disorders) | 6 (7) | 9 (11) | 4 (5) | 8 (11)
Eyelid oedema (Eye disorders) | 7 (8) | 3 (3) | 3 (3) | 7 (7)
Retinal haemorrhage (Eye disorders) | 7 (9) | 6 (6) | 5 (6) | 7 (9)
Retinal tear (Eye disorders) | 2 (2) | 7 (7) | 4 (4) | 1 (1)
Retinal depigmentation (Eye disorders) | 6 (6) | 6 (7) | 6 (6) | 4 (4)
Ocular discomfort (Eye disorders) | 5 (5) | 2 (2) | 4 (4) | 5 (5)
Maculopathy (Eye disorders) | 4 (4) | 5 (6) | 2 (2) | 5 (5)
Vitreous floaters (Eye disorders) | 2 (2) | 5 (6) | 4 (4) | 5 (5)
Ocular hyperaemia (Eye disorders) | 4 (6) | 1 (2) | 3 (3) | 0 (0)
Retinal disorder (Eye disorders) | 3 (3) | 3 (3) | 4 (5) | 2 (3)
Cataract subcapsular (Eye disorders) | 0 (0) | 4 (8) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 2 (3) | 4 (5) | 2 (3) | 2 (4)
Anterior chamber inflammation (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Conjunctival oedema (Eye disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Visual disturbance (Eye disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 3 (4) | 3 (3) | 3 (3)
Conjunctival hyperaemia (Eye disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Corneal disorder (Eye disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 3 (4) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Vitreous disorder (Eye disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Corneal bleeding (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Cataract cortical (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Corneal oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Retinal cyst (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Macular hole (Eye disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Corneal striae (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Retinal degeneration (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (2)
Intraocular pressure increased (Investigations) | 4 (4) | 4 (5) | 6 (6) | 5 (5)
Intraocular pressure decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 5 (6)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — Originally coded to General disorders and administration site conditions
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Originally coded to General disorders and administration site conditions
Retinal oedema (Eye disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days